CLINICAL TRIAL: NCT01447550
Title: Treatment of Thromboangiitis Obliterans (Buerger's Disease) With Bosentan
Brief Title: Treatment of Thromboangiitis Obliterans (Buerguer's Disease) With Bosentan
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Joaquin de Haro, M.D., Treatment of thromboangiitis obliterans (Buergueer´s disease) with Bosentan, Hospital Universitario Getafe
Other Study IDs: Buerger-Bosentan
Record Dates: First submitted 2011-10-05; First posted 2011-10-06 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Thromboangiitis Obliterans
Keywords: Bosentan; Buerguer disease
MeSH Terms: conditions — Thromboangiitis Obliterans | interventions — Bosentan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bosentan: Bosentan
  Interventions: Drug: Bosentan

INTERVENTIONS:
Drug: Bosentan — Bosentan therapy consisted of a month's treatment with 62.5 mg bid orally administered. Dose doubled to 125 mg bid after the first month. The full-dose regimen (125 mg/12h) was maintained for the following months or until total healing fo the ulcers.

SUMMARY:
This study assessed the effectiveness and safety of bosentan when administered to thromboangiitis obliterans (Buerger's disease)patients. A clinical pilot study was designed,included in which patients with ulcer and/or pain at rest were treated with bosentan p.o at a dose of 62,5 mg twice daily during the first month, which each thereafter uptitrated to 125 mg twice daily. Study endpoints were clinical improvement rate, major or minor amputation rate, hemodynamic changes, changes in endothelial function and angiographic changes.

12 patients were included were current smokers. With bosentan treatment, no new ischemic lesions were observed in all but one patient. Overall, clinical improvement was observed in 12 of the 13 extremities (92%). Only two of 13 extremities underwent amputation after bosentan treatment. As assessed by digital arteriography with subtraction or angio-magnetic resonance image an increase of distal flow was observed in 10 out of the 12 patients. All patients experienced a statistically significant improvement in their BAFMD values (means:1.8 at baseline;6.6 at the end of the treatment;12.7 three months after the end of the treatment;p<0.01). In conclusion: Bosentan treatment may result in an improvement of clinical, angiographic, hemodynamic and endothelial function outcome. Bosentan deserves further investigation in the management TAO patients.

ELIGIBILITY:
Inclusion Criteria:

* Critical ischemia in any extremity, causing pain at rest or non-healing ischemic ulcers, present for at least four weeks with no evidence of improvement in response to conventional treatment.

Exclusion Criteria:

* Being candidates for surgical or endovascular revascularisation of the extremity studied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Buerger's disease
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Clinical improvement rate | 4-6 months
  Clinical improvement rate (absence of new throphic lesions, ulcer healing process, pain relief, complete absence of pain), major of minor amputation rate
Clinical improvement rate | 4-6 months
  Clinical improvement rate (abscence of new throphic lesions, ulcer healing process, pain relief, complete absence of pain), major of minor amputation rate
Clinical improvement rate | 4-6 months
  Clinical improvement rate (absence of new throphic lesions, ulcer healing process, pain relief, complete absense of pain), major of minor amputation rate

SECONDARY OUTCOMES:
haemodynamics, endothelial function and angiographic changes | 4-6 months
  Hemodynamic changes as measured by means of ABI, changes in endothelial funtion as measured by means of the brachial artery flow-mediated dilation test (BAFMD) and angiographic changes as measured by means of arteriography with digital substraction or an angio-magnetic resonance image (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin De Haro, MD,PhD, Principal Investigator — Hospital Universitario de Getafe
Locations (2):
- Spain (2):
  - Hospital Universitario de Getafe, Getafe, Getafe
  - Hospital Universitario Getafe, Getafe, Madrid

REFERENCES:
- [Derived] De Haro J, Bleda S, Acin F. An open-label study on long-term outcomes of bosentan for treating ulcers in thromboangiitis obliterans (Buerger's disease). Int J Cardiol. 2014 Dec 15;177(2):529-31. doi: 10.1016/j.ijcard.2014.08.107. Epub 2014 Aug 23. No abstract available. PMID 25217217
- [Derived] De Haro J, Acin F, Bleda S, Varela C, Esparza L. Treatment of thromboangiitis obliterans (Buerger's disease) with bosentan. BMC Cardiovasc Disord. 2012 Feb 14;12:5. doi: 10.1186/1471-2261-12-5. PMID 22333218